CLINICAL TRIAL: NCT03854656
Title: Effect of Time-restricted Eating on Behaviour and Metabolism in Overweight Individuals at High Risk of Type 2 Diabetes - the RESET Study
Brief Title: Effect of Time-restricted Eating on Behaviour and Metabolism in Overweight Individuals at High Risk of Type 2 Diabetes
Acronym: RESET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristine Færch (Other)
Collaborators: University of Copenhagen (Other); Aalborg University Hospital (Other); IMotions A/S (Industry); University of Leeds (Other); Salk Institute for Biological Studies (Other)
Responsible Party: Sponsor-Investigator, Kristine Færch, Senior Researcher and Team Leader, PhD, Steno Diabetes Center Copenhagen
Organization: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NNF17OC0027822
Record Dates: First submitted 2019-02-18; First posted 2019-02-26 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Overweight and Obesity; PreDiabetes
Keywords: Overweight; Obesity; Time-restricted eating; Prediabetes
MeSH Terms: conditions — Overweight; Obesity; Prediabetic State; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control group for 13 weeks (n=50). Participants will receive advice about a healthy lifestyle according to the national dietary recommendations from the Danish Health Authority.
- Time-restricted eating (Experimental): Time-restricted eating for 13 weeks (n=50). In addition to the intervention, participants will receive advice about a healthy lifestyle according to the national dietary recommendations from the Danish Health Authority.
  Interventions: Other: Time-restricted eating

INTERVENTIONS:
Other: Time-restricted eating — Participants will be instructed to eat within a self-selected 10-hour timeframe between 6AM and 8PM every day. All food/beverages except water must be consumed within the time-interval. Staff will help participants select a time-interval that fits into their daily life and optimally fulfil the following guiding principles:
  1. The first food item/beverage of the day should optimally be ingested at least 2 hours after usual wake-up time
  2. The last food item/beverage of the day should optimally be ingested at least 3 hours before usual bed time
  Diet is ad libitum and with no further dietary restrictions. Participants will receive advice about a healthy lifestyle according to the national dietary recommendations from the Danish Health Authority.
  Arms: Time-restricted eating

SUMMARY:
The aim of the present study is to investigate effects of 12 weeks time-restricted eating on behaviour and metabolism in individuals with overweight or obesity at high risk of type 2 diabetes.

DETAILED DESCRIPTION:
Overweight and obese individuals with pre-diabetes or with a family history of diabetes or cardiovascular disease (CVD) are at high risk for developing type 2 diabetes (T2D) and CVD. Current prevention and treatment of obesity and T2D include energy restricted diets and increased levels of physical activity; however, adequate adherence to such strategies is difficult, and maintenance is challenging for most individuals, which stresses the need for feasible and sustainable interventions.

Circadian rhythms of behaviour and metabolism are closely related to the daily light/dark cycle and sleep-wake patterns and timing of food intake and fasting periods may affect the circadian rhythms of metabolic organs. In an evolutionary perspective, the pattern of food consumption has been characterised by periods of caloric intake when food was available and subsequent periods of fasting 9. This cyclic pattern leads to cycles of absorption and storage of energy and utilisation of the energy for e.g. tissue repair, stress resistance and vitality where expression of metabolic regulators coordinates with cellular processes, leading to efficient metabolism 10. Factors including the 24-hour availability of energy-dense foods, busy time schedules, different eating and sleep patterns during weekdays and weekends (i.e. 'social jetlag') challenge the feeding-fasting paradigm. Recent data suggest that an erratic diurnal eating pattern characterised by food intake largely spread throughout hours awake (≥15 h) and a concomitant short fasting period is highly prevalent in humans and animal suggest that circadian misalignment of food intake is associated with adverse metabolic effects. A number of animal studies and a few small studies in humans have reported promising effects of time-restricted eating (TRE), without concomitant dietary restrictions, on body weight and other cardiometabolic risk factors. There is a lack of randomized controlled trials investigating effect of TRE in individuals at high risk of type 2 diabetes and cardiovascular diseases.

The aim of the present study is to investigate effects of 12 weeks TRE on behaviour and metabolism in individuals with overweight or obesity at high risk of type 2 diabetes. Maintenance will be assessed at a follow-up visit 13 weeks after completion of the trial (26 weeks). Testing will be conducted at baseline and after 6, 12, and 26 weeks. Participants are instructed to follow randomization during one week assessment periods after testing at 6 and 12 weeks. Therefore, the total duration of the intervention is 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥30 kg/m2 or BMI ≥25 kg/m2 in combination with pre-diabetes (HbA1c ≥39-<48 mmol/mol)
* Habitual eating/drinking window ≥12 hours (including foods/snacks and energy containing beverages e.g. soft drinks (except of water)) and an eating/drinking window of ≥14 hours minimum one day per week

Exclusion criteria

* Daily smoking
* For women: pregnancy, planned pregnancy (within the study period) or lactating
* Frequent travels over time zones (max one return trip/travel over times zones (˃one hour time difference) during the 13 weeks intervention).
* Shift work or partner engaged in shift work (if it affects the person's sleep and eating pattern)
* Unable to understand the informed consent and the study procedures
* Self-reported history of an eating disorder during the past three years
* Self-reported weight change (>5 kg) within three months prior to inclusion
* Diabetes
* HbA1c ≥48 mmol/mol
* Uncontrolled medical issues including but not limited to cardiovascular pulmonary, rheumatologic, hematologic, oncologic, infectious, gastrointestinal or psychiatric disease; diabetes or other endocrine disease; immunosuppression
* Current treatment with medication or medical devices which significantly affect glucose metabolism, appetite, or energy balance
* Current treatment with antidepressants
* Bariatric surgery
* Implanted or portable electro-mechanical medical device such as a cardiac pacemaker, defibrillator or infusion pump
* Celiac disease, Crohn's disease, ulcerative colitis or proctitis
* Alcohol/drug abuse or in treatment with disulfiram at time of inclusion
* Concomitant participation in other intervention studies
* Not able to eat ≥85% of the test meal because of e.g. allergy

Specific exclusion criteria for participants receiving SmartPillTM (n=60)

* Gastrointestinal symptoms or diseases such as regular (weekly) abdominal pain, dysphagia, gastric bezoars, strictures, fistulas, bowel obstructions or diverticulitis
* Current treatment with medication or medical devices which significantly affect gastrointestinal motility or transit time (prokinetics, antidiarrheals, laxatives, or opioids)
* Gastrointestinal surgery within 3 months before inclusion

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Change in body weight (kg) | Change from baseline to the end of the intervention (after 12 weeks)
  Measured in fasted state on a digital scale

SECONDARY OUTCOMES:
Body weight (kg) | Changes from baseline. Fasted state at all four visits (Baseline and after 6, 12, and 26 weeks)
  Measured on a digital scale
Body mass index (kg/m^2) | Changes from baseline. Fasted state at all four visits (Baseline and after 6, 12, and 26 weeks)
  Calculated from body weight (kg) and height (m)
Fat mass (kg) | Changes from baseline. Fasted state at all four visits (Baseline and after 6, 12, and 26 weeks)
  Measured by Dual-energy X-ray Absorptiometry
Fat free mass (kg) | Changes from baseline. Fasted state at all four visits (Baseline and after 6, 12, and 26 weeks)
  Measured by Dual-energy X-ray Absorptiometry
Fat percentage (%) | Changes from baseline. Fasted state at all four visits (Baseline and after 6, 12, and 26 weeks)
  Measured by Dual-energy X-ray Absorptiometry
Waist circumference (cm) | Changes from baseline. Fasted state at all four visits (Baseline and after 6, 12, and 26 weeks)
  Measured using tape measure
Hip circumference (cm) | Changes from baseline. Fasted state at all four visits (Baseline and after 6, 12, and 26 weeks)
  Measured using tape measure
HbA1c (mmol/mol and %) | Changes from baseline. All four visits (Baseline and after 6, 12, and 26 weeks)
  Assessed from blood samples at all visits
Systolic blood pressure (mmHg) | Changes from baseline. Measured at all four visits (Baseline and after 6, 12, and 26 weeks)
  Measured under resting and fasting conditions
Diastolic blood pressure (mmHg) | Changes from baseline. Measured at all four visits (Baseline and after 6, 12, and 26 weeks)
  Measured under resting and fasting conditions
Heart rate (bpm) | Changes from baseline. Measured at all four visits (Baseline and after 6, 12, and 26 weeks)
  Measured under resting and fasting conditions during measurements of blood pressure and in the supine position by a handheld ECG measuring device (Vagus™)
Resting energy expenditure (kcal/day) | Changes from baseline. Measured at visits at baseline and after 12 weeks
  Measured by indirect calorimetry under resting and fasting conditions
Substrate oxidation (respiratory exchange ratio) | Changes from baseline. Measured at visits at baseline and after 12 weeks
  Measured by indirect calorimetry under resting and fasting conditions
Metabolites | Changes from baseline. Measured in the blood in the fasted state at all four visits (Baseline and after 6, 12, and 26 weeks) and during a mixed meal test (4 hours) at baseline and end of the intervention (after 12 weeks)
  Fasting and postprandial (after a standard mixed breakfast meal) concentrations of metabolites including but not limited to: glucose, lipids, cholesterol, free-fatty acids, and amino acids
Hormones | Changes from baseline. Measured in the blood in the fasted state at all four visits (Baseline and after 6, 12, and 26 weeks) and during a mixed meal test (4 hours) at baseline and end of the intervention (after 12 weeks)
  Fasting and postprandial (after a standard mixed breakfast meal) concentrations of hormones related to regulation of appetite, glucose and lipid metabolism (including but not limited to: insulin, glucagon, ghrelin, glucagon-like peptide-1 (GLP-1), glucose-dependent insulinotropic polypeptide (GIP) and peptide YY (PYY), leptin, fibroblast growth factor 19 (FGF-19), fibroblast growth factor 21 (FGF-21), growth differentiation factor 15 (GDF-15)).
Circulating proteins that associate with low-grade inflammation and lipid metabolism | Changes from baseline. Fasted state at all four visits (Baseline and after 6, 12, and 26 weeks)
  Fasting levels of circulating proteins that associate with low-grade inflammation and lipid metabolism. Such proteins are captured by mass-spectrometry driven analyses of the plasma proteome i.e. proteins circulating in the blood
Respiratory and glycolytic capacities of isolated peripheral blood mononuclear cells (PBMCs) | Changes from baseline. Fasted state at all four visits (Baseline and after 6, 12, and 26 weeks) and during a mixed meal test at baseline and end of the intervention (after 12 weeks)
  Measured using the Seahorse method, which measures mitochondrial respiration
Heart rate response to standing up from the supine position | Changes from baseline. Measured at visits at baseline and end of the intervention (after 12 weeks)
  Measured by a handheld ECG measuring device (Vagus™).
Heart rate response to inhalation and exhalation | Changes from baseline. Measured at visits at baseline and end of the intervention (after 12 weeks)
  Measured by a handheld ECG measuring device (Vagus™).
Heart rate response to forced exhalation during rest (valsalva maneuver) | Changes from baseline. Measured at visits at baseline and end of the intervention (after 12 weeks)
  Measured by a handheld ECG measuring device (Vagus™).
Gastric emptying time (hours and minutes) | Changes from baseline. Time after consumption of the standard mixed meal at baseline and end of the intervention (after 12 weeks).
  Measured using the SmartPill™ technique. The SmartPill™ is ingested together with a standard mixed breakfast meal
Small bowel transit time (hours and minutes) | Changes from baseline. Time after consumption of the standard mixed meal at baseline and end of the intervention (after 12 weeks).
  Measured using the SmartPill™ technique. The SmartPill™ is ingested together with a standard mixed breakfast meal
Large bowel transit time (hours and minutes) | Changes from baseline. Time after consumption of the standard mixed meal at baseline and end of the intervention (after 12 weeks).
  Measured using the SmartPill™ technique. The SmartPill™ is ingested together with a standard mixed breakfast meal
Total gastrointestinal transit time (hours and minutes) | Changes from baseline. Time after consumption of the standard mixed meal at baseline and end of the intervention (after 12 weeks).
  Measured using the SmartPill™ technique. The SmartPill™ is ingested together with a standard mixed breakfast meal
Motility index | Changes from baseline. Time after consumption of the standard mixed meal at baseline and end of the intervention (after 12 weeks).
  Calculated based on amplitudes and number of contractions measured using the SmartPill™ technique. The SmartPill™ is ingested together with a standard mixed breakfast meal
Attention measured using eye tracking | Changes from baseline. Fasted state at all four visits (Baseline and after 6, 12, and 26 weeks) and during a mixed meal test at baseline and end of the intervention (after 12 weeks)
  Eye tracking metrics including gaze duration bias, gaze direction bias, fixations, saccades, pupil size/dilation, distance to screen, ocular vergence and blinks to measure attention in response to looking at food pictures during the computerized Leeds Food Preference Questionnaire
Emotions measured using facial expression analyses | Changes from baseline. Fasted state at all four visits (baseline and after 6, 12, and 26 weeks) and during a mixed meal test at baseline and end of the intervention (after 12 weeks)
  Facial expression analyses using computer-vision algorithms (AFFDEX) to measure emotions in response to looking at food pictures during the computerized Leeds Food Preference Questionnaire
Arousal measured using galvanic skin response | Changes from baseline. Fasted state at all four visits (Baseline and after 6, 12, and 26 weeks) and during a mixed meal test at baseline and end of the intervention (after 12 weeks)
  Changes in conductivity of the skin (galvanic skin response) in response to looking at food pictures during the computerized Leeds Food Preference Questionnaire
Food choice | Changes from baseline. Fasted state at all four visits (Baseline and after 6, 12, and 26 weeks) and during a mixed meal test at baseline and end of the intervention (after 12 weeks)
  Food choice of food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the computerized Leeds Food Preference Questionnaire. Food choice is determined based on frequency of selection made within each food category. The scores range from 0-48 i.e. 0 = foods within a specific food category have not been selected at all to 48 = foods within a specific food category have been selected 48 times
Implicit wanting | Changes from baseline. Fasted state at all four visits (Baseline and after 6, 12, and 26 weeks) and during a mixed meal test at baseline and end of the intervention (after 12 weeks)
  Implicit wanting of food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the computerized Leeds Food Preference Questionnaire. Implicit wanting is assessed based on food choice and response time for selected and non-selected food items as well as mean response time.
Explicit liking | Changes from baseline. Fasted state at all four visits (Baseline and after 6, 12, and 26 weeks) and during a mixed meal test at baseline and end of the intervention (after 12 weeks)
  Explicit liking of 16 food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the computerized Leeds Food Preference Questionnaire. Explicit liking is rated using visual analogue scales and the range is 0-100. Each end represents the extremes e.g. Question: "how pleasant would it be to taste this food right now?" Answer: "not at all" (rated 0 on the 0-100 scale) to "extremely" (rated 100 on the 0-100 scale)
Explicit wanting | Changes from baseline. Fasted state at all four visits (Baseline and after 6, 12, and 26 weeks) and during a mixed meal test at baseline and end of the intervention (after 12 weeks)
  Explicit wanting of 16 food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the computerized Leeds Food Preference Questionnaire. Explicit wanting is rated using visual analogue scales and the range is 0-100. Each end represents the extremes e.g. Question: "how much do you want some of this food now?" Answer: "not at all" (rated 0 on the 0-100 scale) to "extremely" (rated 100 on the 0-100 scale).
Insulin sensitivity (indices) | At all four visits (Baseline and after 6, 12, and 26 weeks)
  Including but not limited to the Matsuda index
Insulin resistance (indices) | At all four visits (Baseline and after 6, 12, and 26 weeks)
  Including but not limited to Homeostaic Model Assessment for Insulin Resistance (HOMA-IR)
Subjective appetite | Changes from baseline. Fasted state at all four visits (Baseline and after 6, 12, and 26 weeks) and during a mixed meal test at baseline and end of the intervention (after 12 weeks)
  Rated using visual analogue scales and includes sensations of: Hunger, fullness, satiety, prospective food consumption, wellbeing, nausea, thirst, desire to eat meat, salty, and sweet. The scale range is 0-100 and each end represent the extremes e.g. hunger rating: "I am not hungry at all" to "I have nerver been this hungry before".
Mean amplitude of glycaemic excursions (MAGE) | Changes from baseline. Measured 7 days after the test days at baseline and after 6 and 12 weeks
  Measured using continous glucose monitoring
Continuous overall net glycaemic action (CONGA) | Changes from baseline. Measured 7 days after the test days at baseline and after 6 and 12 weeks
  Measured using continous glucose monitoring
Daily time spent above different glucose concentrations (e.g. >6.1 mmol/L, >7.0 mmol/L, >7.8 mmol/L, and >11.1 mmol/L) | Changes from baseline. Measured 7 days after the test days at baseline and after 6 and 12 weeks
  Measured using continous glucose monitoring.
Mean glucose concentrations | Changes from baseline. Measured 7 days after the test days at baseline and after 6 and 12 weeks
  Measured using continous glucose monitoring.
Standard deviation of glucose concentrations | Changes from baseline. Measured 7 days after the test days at baseline and after 6 and 12 weeks
  Measured using continous glucose monitoring.
Variation coefficients of glucose concentrations | Changes from baseline. Measured 7 days after the test days at baseline and after 6 and 12 weeks
  Measured using continous glucose monitoring.
Physical activity (time spent at different intensities) | Changes from baseline. Measured 7 days after the test days at baseline and after 6 and 12 weeks
  Sedentary time, light, moderate and vigorous intensity physical activity. Assessed from 24 h/day accelerometry
Physical activity (counts/min) | Changes from baseline. Measured 7 days after the test days at baseline and after 6 and 12 weeks
  Assessed from 24 h/day accelerometry
Physical activity energy expenditure (kcal/day) | Changes from baseline. Measured 7 days after the test days at baseline and after 6 and 12 weeks
  Assessed from 24 h/day accelerometry
Physical activity (MET hours) | Changes from baseline. Measured 7 days after the test days at baseline and after 6 and 12 weeks
  Assessed from 24 h/day accelerometry
Timing of physical activity (hh:mm) | Changes from baseline. Measured 7 days after the test days at baseline and after 6 and 12 weeks
  Assessed from activity logs and 24 h/day accelerometry
Energy intake (kcal/day) | Changes from baseline. Registered 3 days after the test days at baseline and after 6 and 12 weeks
  Assessed from diet records
Macronutrient intake (energy percentage) | Changes from baseline. Registered 3 days after the test days at baseline and after 6 and 12 weeks
  Assessed from diet records
Timing of dietary intake (hh:mm) | Changes from baseline. Registered 3 days after the test days at baseline and after 6 and 12 weeks
  Assessed from diet records
Sleep timing (hh:mm) | Changes from baseline. Registered and measured for 7 days after the test days at baseline and after 6 and 12 weeks
  Including bedtime, sleep onset, wake-up, time out of bed, sleep midpoint. Assessed from sleep logs and 24 h/day accelerometry
Sleep duration (min) | Changes from baseline. Registered and measured for 7 days after the test days at baseline and after 6 and 12 weeks
  Assessed from sleep logs and 24 h/day accelerometry
Sleep variability (min) | Changes from baseline. Registered and measured for 7 days after the test days at baseline and after 6 and 12 weeks
  Variability in bedtime, wake-up, sleep duration and sleep midpoint. Assessed from sleep logs and 24 h/day accelerometry
Sleep onset latency (min) | Changes from baseline. Registered and measured for 7 days after the test days at baseline and after 6 and 12 weeks
  Assessed from sleep logs and 24 h/day accelerometry
Sleep efficiency (%) | Changes from baseline. Measured for 7 days after the test days at baseline and after 6 and 12 weeks
  Assessed from 24 h/day accelerometry
Wakefulness (min) | Changes from baseline. Measured for 7 days after the test days at baseline and after 6 and 12 weeks
  Assessed from 24 h/day accelerometry
Self-reported gastrointestinal symptoms (part 1) | Changes from baseline. Assessed at all four visits (Baseline and after 6, 12, and 26 weeks)
  Assessed from the questionnaires the Gastrointestinal Symptom Rating Scale (GSRS). Rated on 7-point likert scales. Range: 1 = absence of symptoms to 7 = very severe symptoms.
Self-reported gastrointestinal symptoms (part 2) | Changes from baseline. Assessed at all four visits (Baseline and after 6, 12, and 26 weeks)
  Assessed from the Gastrointestinal Symptom Score (PAGI-SYM). Rated on 6-point likert scales. Range: 1 = absence of symptoms to 6 = very severe symptoms.
Self-reported gastrointestinal symptoms (part 3) | Changes from baseline. Registered 7 days after the test days at baseline and after 12 weeks
  Number of symptoms. Assessed from logs.
Self-reported autonomic symptoms | Changes from baseline. Assessed at all four visits (Baseline and after 6, 12, and 26 weeks)
  Assessed from the questionnaire COMPASS31
Self-reported control over eating | Changes from baseline. Assessed at all four visits (Baseline and after 6, 12, and 26 weeks)
  Assessed from the questionnaire Control over Eating Questionnaire
Self-reported sleepiness | Changes from baseline. Assessed at all four visits (Baseline and after 6, 12, and 26 weeks)
  Assessed from the questionnaire the Epworth Sleepiness Scale
Self-reported sleep quality | Changes from baseline. Assessed at all four visits (Baseline and after 6, 12, and 26 weeks)
  Assessed from the questionnaire Pittsburgh Sleep Quality Index
Self-reported chronotype | Changes from baseline. Assessed at all four visits (Baseline and after 6, 12, and 26 weeks)
  Assessed from the Munich Chronotype Questionnaire
Self-reported physical activity | Changes from baseline. Assessed at all four visits (Baseline and after 6, 12, and 26 weeks)
  Assessed from questionnaire International Physical Activity Questionnaire
Self-reported overall health and wellbeing | Changes from baseline. Assessed at all four visits (Baseline and after 6, 12, and 26 weeks)
  Assessed from the questionnaire Self-reported health (SF-36 health survey)
Self-reported eating behavior | Changes from baseline. Assessed at all four visits (Baseline and after 6, 12, and 26 weeks)
  Assessed from The Dutch Eating Behavior Questionnaire
Self-reported night eating | Changes from baseline. Assessed at all four visits (Baseline and after 6, 12, and 26 weeks)
  Assessed from The Night Eating Questionnaire
Daily eating/drinking window (hh:min) | Registrered every day (13 weeks intervention and 13 weeks follow-up period)
  Time of first and last meal/beverage
Microbiome content and diversity | Changes from baseline. Collected before or during test days at visits at baseline and after 12 weeks
  Determined from stool samples. Bacterial DNA and RNA will be purified from the stool samples and changes in the microbiome composition and function will be estimated based on sequencing of the microbiomes' DNA and RNA. Includes but is not limited to the Firmicute/Bacteroidete ratio.
Motivation for participation (qualitative methods) | Visits at baseline and after 12 and 26 weeks. Potential drop-outs will be interviewed at the specific time point.
  Themes and aspects related to motivation for participation will be assessed based on interviews with the participants including completers and potential drop-outs.
Feasibility of the intervention (qualitative methods) | Visits at baseline and after 12 and 26 weeks. Potential drop-outs will be interviewed at the specific time point.
  Themes and aspects related to feasibility of the intervention will be assessed based on interviews with the participants including completers and potential drop-outs.
Satisfaction with the intervention (qualitative methods) | Visits at baseline and after 12 and 26 weeks. Potential drop-outs will be interviewed at the specific time point.
  Themes and aspects related to satisfaction with the intervention will be assessed based on interviews with the participants including completers and potential drop-outs.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Færch, PhD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quist JS, Pedersen HE, Jensen MM, Clemmensen KKB, Bjerre N, Ekblond TS, Uldal S, Storling J, Wewer Albrechtsen NJ, Holst JJ, Torekov SS, Nyeland ME, Vistisen D, Jorgensen ME, Panda S, Brock C, Finlayson G, Blond MB, Faerch K. Effects of 3 months of 10-h per-day time-restricted eating and 3 months of follow-up on bodyweight and cardiometabolic health in Danish individuals at high risk of type 2 diabetes: the RESET single-centre, parallel, superiority, open-label, randomised controlled trial. Lancet Healthy Longev. 2024 May;5(5):e314-e325. doi: 10.1016/S2666-7568(24)00028-X. Epub 2024 Apr 5. PMID 38588687
- [Derived] Jensen MM, Pedersen HE, Clemmensen KKB, Ekblond TS, Ried-Larsen M, Faerch K, Brock C, Quist JS. Associations Between Physical Activity and Gastrointestinal Transit Times in People with Normal Weight, Overweight, and Obesity. J Nutr. 2024 Jan;154(1):41-48. doi: 10.1016/j.tjnut.2023.06.005. Epub 2023 Jun 12. PMID 37315794
- [Derived] Quist JS, Jensen MM, Clemmensen KKB, Pedersen H, Bjerre N, Storling J, Blond MB, Wewer Albrechtsen NJ, Holst JJ, Torekov SS, Vistisen D, Jorgensen ME, Panda S, Brock C, Finlayson G, Faerch K. Protocol for a single-centre, parallel-group, randomised, controlled, superiority trial on the effects of time-restricted eating on body weight, behaviour and metabolism in individuals at high risk of type 2 diabetes: the REStricted Eating Time (RESET) study. BMJ Open. 2020 Aug 26;10(8):e037166. doi: 10.1136/bmjopen-2020-037166. PMID 32847912

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT03854656/SAP_000.pdf